CLINICAL TRIAL: NCT02555202
Title: Validation of the French Version of the London Chest Activity of Daily Living Scale (LCADL) and the Dyspnea-12 Questionnaire
Brief Title: Validation of French Version of LCADL and Dyspnea-12
Acronym: LCADL
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: LCADL (RB 15.037)
Record Dates: First submitted 2015-09-16; First posted 2015-09-21 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2016-09

CONDITIONS: Copd
Keywords: dyspnea
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The main objective of this study is to develop and to validate a French version of the London Chest Activity of Daily Living (LCADL) and the Dyspnea 12 and to determine the reliability of this version for the evaluation of the dyspnea in the Activity of Daily Living in COPD patients (stages severe and very severe).

ELIGIBILITY:
Inclusion Criteria:

* COPD with FEV1< 50% of predictive value

Exclusion Criteria:

* FEV1> 50% of predictive value
* Patients with an exacerbation of COPD in the previous 30 days the inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: copd patients stage 3 and 4
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2015-10-15 (Actual); Primary Completion 2016-09-30 (Actual); Study Completion 2016-09-30 (Actual)

PRIMARY OUTCOMES:
the Saint-Georges questionnaire, item Activity | 15 days
  by comparison with item activities of the Saint-Georges questionnaire for the LCADL
MMRC Dyspnea scale | 15 days
  by comparison with MMRC dyspnea scale for the dyspnea 12

CONTACTS AND LOCATIONS:
Overall Officials: Francis Couturaud, MD,PhD, Principal Investigator — CHU BREST, Département de médecine interne et pneumologie EA 3878, CIC INSERM 1412, IFR 148
Locations (1):
- Brest University hospital, Morlaix, France